CLINICAL TRIAL: NCT01708421
Title: Phenotypic and Genotypic Associations With Symptom Clusters During Childhood Leukemia Treatment
Brief Title: Symptom Clusters in Children With Leukemia
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00037891
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Childhood Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A baseline CSF sample will be obtained prior to intrathecal chemotherapy. CSF biomarkers will be obtained at the initiation of post-induction, 4 and 6 months into post-induction therapy, and at the start of maintenance therapy.A saliva sample will be obtained for genotypic analysis at one of the four data collection times.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to examine the phenotypic and genotypic characteristics and their associations with symptom clusters experienced during treatment for childhood leukemia.

DETAILED DESCRIPTION:
A repeated measures research design will evaluate phenotypic and genotypic treatment-related symptom associations experienced by children and adolescents 3-17 years of age with a diagnosis of leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Phenotypic and genotypic treatment-related symptom associations will be evaluated in children and adolescents 3-18 years of age with a diagnosis of leukemia.

Exclusion Criteria:

* Children without a definite diagnosis of leukemia will be excluded.
* Children must be able to understand and answer the questions on the questionnaires.
* Children with have a cognitive impairment (e.g. Down syndrome) will not be able to complete the questionnaires and will not be eligible for the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between 3-18 years of age undergoing treatment for leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2012-11; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Hockenberyy, PhD, Principal Investigator — Duke University School of Nursing
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - Children's Hospitals & Clinics of Minnesota, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine/ Texas Children's Cancer Center, Houston, Texas